CLINICAL TRIAL: NCT01809886
Title: Reversal With Sugammadex (BRIDION ®) From Deep Neuromuscular Blockade Induced by Rocuronium in Children: Randomised Clinical Trial of Efficacy and Safety
Brief Title: Reversal With Sugammadex From Deep Neuromuscular Blockade Induced by Rocuronium in Children: Randomised Clinical Trial
Acronym: SUGAPED-01
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fundacion para la Formacion e Investigacion Sanitarias de la Region de Murcia (Other)
Collaborators: Hospital Universitario Virgen de la Arrixaca (Other); Hospital Universitario Santa Maria del Rosell (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT-PED-2010-01CT; 2011-000401-50 (EudraCT Number)
Record Dates: First submitted 2012-08-28; First posted 2013-03-13 (Estimated); Last update posted 2014-03-06 (Estimated); Status verified 2014-03

CONDITIONS: Neuromuscular Blockade
Keywords: Neuromuscular relaxants; short-term pediatric surgery; reverses neuromuscular blockade
MeSH Terms: interventions — Sugammadex; Neostigmine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sugammadex (Experimental): 50 patients, aged between 2 and 11 years scheduled for surgery and requiring muscle relaxation. The reversal will be made with sugammadex 4 mg/kg when surgery is over, maintaining a profound block level until that point in time (no response to TOF and PTC<2).
  Interventions: Drug: Sugammadex
- Neostigmina (Active Comparator): 50 patients aged between 2 and 11 years scheduled for surgery and requiring muscle relaxation. The reversal will be made with neostigmine 0. 05 mg/kg and atropine 0.025 mg/kg (conventional reverser treatment) when surgery is over, maintaining a profound block level unit that point in time (no response to TOF and PTC<2).
  Interventions: Drug: Neostigmine

INTERVENTIONS:
Drug: Sugammadex — 50 patients, aged between 2 and 11 years scheduled for surgery and requiring muscle relaxation. The reversal will be made with sugammadex 4 mg/kg when surgery is over, maintaining a profound block level until that point in time (no response to TOF and PTC<2).
  Arms: Sugammadex
Drug: Neostigmine — 50 patients aged between 2 and 11 years scheduled for surgery and requiring muscle relaxation. The reversal will be made with neostigmine 0. 05 mg/kg and atropine 0.025 mg/kg (conventional reverser treatment) when surgery is over, maintaining a profound block level unit that point in time (no response to TOF and PTC<2).
  Arms: Neostigmina

SUMMARY:
The purpose of this clinical trial is to prove that the administration of sugammadex at a dose of 4 mg/kg for counteracting deep blockage [without train-of-four (TOF) ratio response and post-tetanic count (PTC) < of 2 induced and maintained with Rocuronium in pediatric patients for short-term elective surgery.

DETAILED DESCRIPTION:
Muscle relaxing facilitates endotracheal intubation and surgical access. Muscle relaxants have a long duration with the possibility of residual muscle relaxation after surgery (over 40% of patients), and ventilatory problems (hypoxia, hypercapnia, atelectasis, airway collapse) that raise postoperative morbidity and mortality.

All of these facts are accentuated in the pediatric patient due to the reduced airway caliber which tends lead to obstruction and bronchospasm. So far, the effect of muscle relaxants has only been partially reversed by anticholinesterase (neostigmine), which has the limitation of its short duration of action (8-9 minutes) and has many side effects (bradycardia, hypotension, increased salivation, vomiting, dyspnea and bronchoconstriction). It also needs to be combined with anticholinergic (atropine), which causes a dry mouth, blurred vision and tachycardia.

At present, the introduction of sugammadex (Bridion®), an antagonist of nondepolarizing the neuromuscular relaxant rocuronium, may lead to an extraordinary breakthrough. It is the only antagonist able to encapsulate and fully eliminate the muscle relaxant to avoid residual effects and respiratory complications. Muscle strength can be retrieved at any time, without waiting for relaxant metabolism (30 to 40 minutes) and without using the usual classical antidotes (neostigmine and atropine), which produce many undesirable effects that become more troublesome in the postoperatory phase. Sugammadex lacks intrinsic activity and is considered safe, without significant side effects and can be used in cardiovascular or respiratory diseases.

ELIGIBILITY:
Inclusion Criteria:

* Children of both sexes,
* Aged between two and eleven years who have undergone surgery for procedures of short duration (less than one hour) and requiring muscle relaxation.
* Informed consent signed by parents or guardians

Exclusion Criteria:

* No signed informed consent by parent/guardian,
* Anticipated difficult airway,
* Neuromuscular disease,
* Liver and/or renal failure,
* Personal or family history of malignant hyperthermia,
* Previous allergic reaction to any anesthetic.
* Treated at the time of the study with aminoglycosides, magnesium, or anticonvulsants.

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2011-10; Primary Completion 2013-10 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
The time in seconds which has elapsed until a T4/T1 ratio >0,9. | After surgery (Up to 10 h)

SECONDARY OUTCOMES:
Heart Rate (beats / min) | After surgery (Up to 10 h)
Systolic and Diastolic blood pressure (mm HG) | After surgery (up to 10 h)
Arterial oxygen saturation (%) | After surgery (up to 10 h)
Total dose of rocuronium (mg/kg) | After surgery (up to 10 h)
Number of participants with at least One Adverse event (AE) | up to 24 h
Time in seconds from the initial dose administered of rocuronium until the maximum block is achieved(Onset time) | During peri-anesthetic period (up to 10 h)
The time in seconds which has elapsed until a T4/T1 >0,8 is achieved. | After surgery (up to 10 h)
The time in seconds which has elapsed until a T4/T1 ratio >0,7 | After surgery (up to 10 h)

CONTACTS AND LOCATIONS:
Overall Officials: MºDolores Cárceles Barón, MD,PhD, Principal Investigator — Hospital Universitario Virgen de la Arrixaca
Locations (1):
- Mª Dolores Cárceles Barón, El Palmar, Murcia, Spain